CLINICAL TRIAL: NCT00323869
Title: Phase II Trial of Bevacizumab in Combination With Gemcitabine and Carboplatin in Patients With Newly Diagnosed Non-Small Cell Lung Cancer (Excluding Squamous Cell Carcinoma)
Brief Title: Phase II Bevacizumab, Gemcitabine and Carboplatin in Newly Diagnosed Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Eli Lilly and Company (Industry); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Heather Wakelee, Associate Professor of Medicine (Oncology), Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-03730; 96655 (Other: Stanford IRB alternate number); AVF3576s; LUN0013 (Other: OnCore); NCT00323869 (Other: NCT number)
Record Dates: First submitted 2006-05-08; First posted 2006-05-10 (Estimated); Results first posted 2016-07-27 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer; Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Cetuximab; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab + carboplatin + gemcitabine (Experimental): Bevacizumab in combination with carboplatin and gemcitabine:
  •Carboplatin, administered IV at area under the curve (AUC) of 5, every 3 weeks on day 1 of each 3-week cycle (once per cycle) for up to 6 cycles.
  Carboplatin was administered before the gemcitabine infusion:
  •Gemcitabine, administered 1000 mg/m² IV on days 1 and 8 of each 3-week cycle (twice per cycle) for up to 6 cycles
  Bevacizumab was administered 1 hour after end of all chemotherapy infusions:
  •Bevacizumab was administered 15 mg/kg IV on day 1 of each 3-week cycle (once per cycle) for up to 6 cycles in combination with chemotherapy, then continuing until evidence of progressive disease or significant treatment-related toxicity
  Interventions: Drug: Bevacizumab; Drug: Gemcitabine; Drug: Carboplatin

INTERVENTIONS:
Drug: Bevacizumab — Murine humanized anti-vascular endothelial growth factor A (VEGF-A) monoclonal antibody
  Other Names: Avastin; C225; rhuMAb-VEGF
Drug: Gemcitabine — Nucleoside analog
  Other Names: Gemzar
Drug: Carboplatin — Alkylating agent
  Other Names: Paraplatin; CBDCA

SUMMARY:
A multi-center study of bevacizumab in combination with gemcitabine and carboplatin as treatment for newly-diagnosed advanced non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This is a open-label, phase 2, single-arm, multi-center study of bevacizumab combined with gemcitabine and carboplatin. This treatment is for newly-diagnosed advanced non-small cell lung cancer (NSCLC), excluding squamous cell carcinoma. All subjects will receive 15 mg/kg bevacizumab every 3 weeks cycle, 1000 mg/m² of gemcitabine on day 1 and 8 every 3 weeks cycle and carboplatin (AUC= 5 ) every 3 weeks. Carboplasm will be administered 1 hour prior to the gemcitabine infusion, bevacizumab will be administered 1 hour following chemotherapy infusion.

Subjects will receive a maximum of 6 cycles of chemotherapy, but treatment with bevacizumab may continue as long as patients have no evidence of progressive disease and no significant treatment-related toxicities.

ELIGIBILITY:
Inclusion Criteria :

* Age 18 or higher
* Life expectancy of at least 3 months
* ECOG Performance status 0 to 1
* Advanced stage non-small cell lung cancer, NSCLC, Stage IIIB with malignant pleural effusion or Stage 4, excluding squamous cell histology, with measurable or evaluable disease
* No prior systemic therapy for advanced NSCLC (prior therapy for early stage disease with one regimen is acceptable if it was completed at least 6 months prior to study entry)
* Palliative radiotherapy to painful bony metastases is permitted prior to study entry if completed prior to initiation of study treatment, and there are no residual sequelae of therapy such as bone marrow suppression
* Willingness to use appropriate contraception to avoid pregnancy during the study
* Leukocytes ≥ 3,000/µL
* Absolute neutrophil count ≥ 1,500/ µL
* Platelets ≥ 100,000/ µL
* Total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) ≤ 2.5 x institutional upper limit of normal
* Creatinine: Within normal institutional limits
* Creatinine clearance ≥ 60 mL/min/1.73 m² for patients with creatinine levels above institutional normal
* Ability to sign informed consent

Exclusion Criteria:

* Prior systemic treatment for advanced NSCLC (one prior regimen of up to 4 cycles of neoadjuvant or adjuvant therapy for early stage disease will be allowed, if completed at least 6 months prior to study entry)
* Known brain metastases
* Prior treatment with bevacizumab
* History of allergic reactions
* Sensitivity attributed to compounds of similar chemical or biologic composition to bevacizumab
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in any other experimental drug study
* Concomitant chemotherapy, radiotherapy, or investigational agents
* Evidence of bleeding diathesis
* Coagulopathy
* Use of anti-coagulant agents including warfarin, heparin, aspirin, NSAIDs
* Pregnant
* Lactating
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, anticipation of need for major surgical procedure during the course of the study
* Minor surgical procedures within 7 days prior to day 0
* Fine needle aspirations within 7 days prior to day 0
* Core biopsies within 7 days prior to day 0
* Urine protein: creatinine ratio ≥ 1.0 at screening
* History of abdominal fistula within 6 months prior to Day 0
* Gastrointestinal perforation within 6 months prior to Day 0
* Intra-abdominal abscess within 6 months prior to Day 0
* Serious, non-healing wound
* Ulcer
* Bone fracture
* Lung carcinoma of squamous cell histology
* Any histology in close proximity to a major vessel
* Significant cavitation as assessed by treating investigator in consultation with an attending radiologist
* History of hemoptysis (bright red blood of 1/2 teaspoon or more)
* Blood pressure of > 150/100 mmHg
* Unstable angina
* New York Heart Association (NYHA) Grade 2 or greater congestive heart failure
* History of myocardial infarction within 6 months
* History of stroke within 6 months
* Clinically significant peripheral vascular disease
* Psychiatric illness/social situations that would limit compliance with study requirements
* Another active malignancy except for non-melanoma skin cancers
* Inability to comply with study and/or follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather A Wakelee, MD, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - VA Palo Alto Healthcare System, Palo Alto, California
  - Santa Clara Valley Medical Center, San Jose, California
  - Stanford University School of Medicine, Stanford, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Clement-Duchene C, Krupitskaya Y, Ganjoo K, Lavori P, McMillan A, Kumar A, Zhao G, Padda S, Zhou L, Pedro-Salcedo MS, Colevas AD, Wakelee HA. A phase II first-line study of gemcitabine, carboplatin, and bevacizumab in advanced stage nonsquamous non-small cell lung cancer. J Thorac Oncol. 2010 Nov;5(11):1821-5. doi: 10.1097/JTO.0b013e3181f1d23c. PMID 20881641

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab + Carboplatin + Gemcitabine: Bevacizumab in combination with carboplatin and gemcitabine
  Bevacizumab was administered 15 mg/kg IV on day 1 of each 3-week cycle (once per cycle) for up to 6 cycles in combination with chemotherapy, then continuing until evidence of progressive disease or significant treatment-related toxicity Gemcitabine, administered 1000 mg/m2 IV on days 1 and 8 of each 3-week cycle (twice per cycle) for up to 6 cycles Carboplatin, administered IV at area under the curve (AUC) of 5, every 3 weeks on day 1 of each 3-week cycle (once per cycle) for up to 6 cycles
  Carboplatin was administered before gemcitabine infusion.
  Bevacizumab was administered 1 hour after end of all chemotherapy infusions.
  Bevacizumab: Murine humanized anti-vascular endothelial growth factor A (VEGF-A) monoclonal antibody
  Gemcitabine: Nucleoside analog
  Carboplatin: Alkylating agent
Period: Overall Study
Arm/Group | Bevacizumab + Carboplatin + Gemcitabine
Started | 48 (Enrollment)
Treatment Initiation | 47 (One participant died before receiving therapy, not included in analysis)
Completed | 47
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Groups:
- Bevacizumab + Carboplatin + Gemcitabine: Treatment provided in 3-week cycles:
  * 15 mg/kg bevacizumab Day 1 of each cycle
  * 1000 mg/m2 gemcitabine Days 1 and 8 of each cycle
  * Carboplatin (AUC of 5 every 3 weeks)
Arm/Group | Bevacizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 47
Age, Continuous [Mean (Full Range); unit: years] | 59 [35 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 29
  More than one race | 0
  Unknown or Not Reported | 4
Eastern Cooperative Oncology Group (ECOG) performance status [Number; unit: participants] — ECOG performance status
  * 0 = Fully active, able to carry on all pre-disease performance without restriction
  * 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, eg, light house work, office work
  * 2 = Unable to work, must sit or lie > 50% waking hours
  * 3 = Capable of limited selfcare; confined to bed or chair > 50% waking hours
  * 4 = Completely disabled; cannot carry on any selfcare; totally confined to bed/chair
  * 5 = Deceased
  participants
    ECOG 0 | 3
    ECOG 1 | 44
Smoking Status [Number; unit: participants] — Smoking status based on self-declaration between:
  * Never a smoker (< 100 cigarettes in lifetime)
  * Quit and not currently a smoker
  * Currently a smoker.
  participants
    Never a smoker | 19
    Has stopped smoking (ex-smoker) | 7
    Currently a smoker | 21
Non-small Cell Lung Cancer (NSCLC) Histology [Number; unit: participants]
  Adenocarcinoma | 30
  Bronchioloalveolar carcinoma (BAC) | 4
  NSCLC not otherwise specified | 13
Non-small Cell Lung Cancer Stage [Number; unit: participants] — During the time of the trial patients with a malignant pleural effusion as only site of metastases were considered stage III-B (AJCC 6th edition). They were treated the same as stage IV (metastatic). Thus all patients included in this trial had advanced stage NSCLC and if staged under current staging criteria (AJCC 7th edition) all would be considered stage IV (metastatic).
  participants
    NSCLC Stage III-B | 8
    NSCLC Stage IV | 39

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Median progression-free survival (PFS) was assessed as the time to disease progression; toxicity requiring treatment discontinuation; or death.
Time Frame: 18 months
Population: Includes all subjects who initiated treatment
Measure: Median (Full Range); unit: months
Arm/Group | Bevacizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 47
months | 8.7 [7.8 to 17.9]

2. Secondary Outcome: Response Rate (CR + PR + SD)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions, by computed tomography (CT); bone scan; positron emission tomography (PET) scan; and/or magnetic resonance imaging (MRI) as necessary to assess diseasE
  Response determined as the number of subjects with any clinical response (CR + PR + SD) per RECIST criteria.
  * Complete Response (CR) = disappearance of all target lesions
  * Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions
  * Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, or appearance of new cancer lesions
  * Stable Disease (SD): No significant effect, does not meet criteria for PR or PD.
Time Frame: 6 weeks
Population: Includes all subjects who initiated treatment
Measure: Number; unit: participants
Arm/Group | Bevacizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 47
participants | 41

3. Secondary Outcome: Overall Survival (OS)
Description: To evaluate the safety of the combination regimen.
Time Frame: 36 months
Population: Includes all subjects who initiated treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 47
months | 12.8 [10.0 to 16.5]

4. Secondary Outcome: Partial Response (PR)
Description: Number of subjects with PR per RECIST criteria
Time Frame: 6 weeks
Population: Includes all subjects who initiated treatment
Measure: Number; unit: participants
Arm/Group | Bevacizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 47
participants | 7

5. Secondary Outcome: Complete Response (CR)
Description: Number of subjects with CR per RECIST criteria
Time Frame: 6 weeks
Population: Includes all subjects who initiated treatment
Measure: Number; unit: participants
Arm/Group | Bevacizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 47
participants | 0

6. Secondary Outcome: Stable Disease (SD)
Description: Number of subjects with SD per RECIST criteria
Time Frame: 6 weeks
Population: Includes all subjects who initiated treatment
Measure: Number; unit: participants
Arm/Group | Bevacizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 47
participants | 34

7. Secondary Outcome: Time-to-First Event
Description: Median time-to-first event, with events defined as disease progression, death, or toxicity requiring drug discontinuation
Time Frame: 18 months
Population: Includes all subjects who initiated treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 47
months | 6.4 [4.8 to 7.9]

8. Secondary Outcome: Overall Survival (OS) at 12 Months
Description: Number of subjects surviving 1 year after treatment initiation
Time Frame: 12 months
Population: Includes all subjects who initiated treatment
Measure: Number; unit: participants
Arm/Group | Bevacizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 47
participants | 27

9. Secondary Outcome: Overall Survival (OS) at 24 Months
Description: Number of subjects surviving 2 years after treatment initiation
Time Frame: 24 months
Population: Includes all subjects who initiated treatment
Measure: Number; unit: participants
Arm/Group | Bevacizumab + Carboplatin + Gemcitabine
Number analyzed (Participants) | 47
participants | 5

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: All assessments were taken after every two cycles. Evaluations were taken the first 6 weeks, then every 3 weeks
Arm/Group | Bevacizumab + Carboplatin + Gemcitabine
Serious Adverse Events (participants affected / at risk) | 28/47
Other Adverse Events (participants affected / at risk) | 17/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab + Carboplatin + Gemcitabine (N=47)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Death (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hemorrahage (Blood and lymphatic system disorders) | 1 (1) — Nose
Platetes (Blood and lymphatic system disorders) | 1 (1)
Hypotension (Blood and lymphatic system disorders) | 1 (1)
Leukocytes (Blood and lymphatic system disorders) | 1 (1)
Hyponatreamia due to SIADH (Metabolism and nutrition disorders) | 1 (1) — SIADH- syndrome of inappropriate antidiuretic hormone
Pain (General disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Possible Pneumonia
Bilirubin (Metabolism and nutrition disorders) | 1 (1) — hyperbilirubinemia
Hematoma (Blood and lymphatic system disorders) | 1 (1) — Liver Hemorrhage
Pulmonary Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab + Carboplatin + Gemcitabine (N=47)
Neutropenia (Blood and lymphatic system disorders) | 4 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Confusion (Nervous system disorders) | 2 (2)
Leukocytes (Blood and lymphatic system disorders) | 3 (3)
Transaminitis (Metabolism and nutrition disorders) | 1 (1)
Pain (Cardiac disorders) | 1 (1) — Chest
Neutrophilis/Granolocytes (Blood and lymphatic system disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Creatinine (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No